CLINICAL TRIAL: NCT03525431
Title: Genomic Sequencing to Aid Diagnosis in Pediatric and Prenatal Practice: Examining Clinical Utility, Ethical Implications, Payer Coverage, and Data Integration in a Diverse Population.
Brief Title: Clinical Utility of Pediatric Whole Exome Sequencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1U01HG009599-01 (NIH); U01HG009599 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-05-15 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Encephalopathy; Birth Defect; Intellectual Disability; Multiple Congenital Anomaly; Metabolic Disease; Epilepsy; Neuro-Degenerative Disease; Cerebral Palsy; Developmental Delay; Developmental Defect
Keywords: Exome; Sequencing; Clinical Utility; Pediatric; Underrepresented; Underserved
MeSH Terms: conditions — Brain Diseases; Congenital Abnormalities; Intellectual Disability; Abnormalities, Multiple; Metabolic Diseases; Epilepsy; Cerebral Palsy; Learning Disabilities | interventions — Exome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Whole Exome Sequencing (Experimental): Following consent and collection of standardized phenotypic data, probands and biological parents will undergo WES with variant analysis conducted utilizing primary gene lists based on referring clinical indication. After results provision and follow up 6-12 months later, clinical utility will be assessed in those with a positive result (pathogenic or likely pathogenic variant) and those with negative results (no variant returned or a VUS) using specific outcomes at each site to examine effectiveness for both the child and family.
  Interventions: Diagnostic Test: Whole Exome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole Exome Sequencing — Whole Exome Sequencing is a form of Next Generation Sequencing allowing investigators to assess the coding regions of many thousands of genes to find variants implicated in disease.
  Other Names: Next Generation Sequencing

SUMMARY:
The investigator aims to examine the clinical utility of WES, including assessment of a variety of clinical outcomes in undiagnosed pediatric cases.

DETAILED DESCRIPTION:
Next-generation sequencing (NGS) is changing the paradigm of clinical genetic testing. Unlike highly focused single-gene tests, NGS allows one to examine gene panels, the exome, and the whole genome. With the broad array of molecular tests now available, ordering physicians face the conundrum of selecting the best diagnostic tool for patients with suspected genetic conditions. Single-gene testing is often most appropriate for conditions with distinctive clinical features and minimal locus heterogeneity. NGS-based gene panel testing, which can be complemented with chromosomal microarray analysis (CMA) and other ancillary methods, provides a comprehensive and feasible approach for well documented but genetically heterogeneous disorders. Whole exome sequencing (WES) and whole genome sequencing (WGS) have the advantage of enabling parallel interrogation of most of the genes in the human genome. To some, WES is preferable to previously used methods due to higher diagnostic yield, shorter time to diagnosis, and improved cost-efficiency.

The ability to survey the exome opens up both new opportunities and new challenges. For example, all coding regions of known genes must be analyzed when applying WES to undiagnosed cases with unclear inheritance patterns. Current limitations on variant interpretation capabilities and clinical validity raise questions about the clinical utility of WES as either a stand-alone or a first-choice diagnostic test. Additional challenges include pre- and post-test counseling with appropriate and robust informed consent, bioinformatics analysis setup and validation, variant interpretation and classification, the need for policies and protocols concerning the discovery and reporting of secondary findings unrelated to the presenting indication, a requirement for validation of WES results, assurance of conformation to quality control standards, data storage and accessibility, and reimbursement issues.

Introducing WES into pediatric clinical care of underrepresented populations raises additional issues and considerations of payment coverage, access, and standards of care. Beyond the sheer complexity of the test and its results, clinicians and health systems must address numerous considerations, including: private and public insurance coverage; language and culture differences and their implications for genetic counseling and clinician-patient relationships; ability to access follow-up testing and clinical care; and ability to access appropriate treatment and services. These issues and others will affect not only patients' decision-making regarding WES, but also their post-test needs for patient follow up. The importance of systematically assessing the clinical utility of NGS is critical for determining in which clinical and health care contexts WES will be useful and for commencing research on these considerations.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting clinical features suggestive of a genetic etiology, including intellectual disability, seizures, multiple congenital anomalies, metabolic conditions, and neurodegenerative conditions or idiopathic cerebral palsy.
2. A minimum of one biological parent is available and willing to provide a specimen for WES, with a preference for two available parents. At least one parent consenting to WES of the child.

4. Pediatric patients must have had at least one prior genetics appointment or evaluation 5. Pediatric patients may have had a single nucleotide polymorphism (SNP) array or oligonucleotide array that did not provide a diagnosis.

Even though this study is for pediatric patients, maximum age limit was increased to 25, if patients fulfilling the above criteria were being followed by Pediatrics Department since they were younger than 18.

Exclusion Criteria:

1. Prior WES performed for a clinical or research indication
2. Lack of phenotypic indication of a likely underlying genetic etiology
3. Both biological parents are unavailable.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 529 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pui-Yan Kwok, MD/PhD, Principal Investigator — University of California, San Francisco; Barbara Koenig, PhD, Principal Investigator — University of California, San Francisco; Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF Fresno, Fresno, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Benioff Children's Hospital Mission Bay, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Muzny DM, Reid JG, Bainbridge MN, Willis A, Ward PA, Braxton A, Beuten J, Xia F, Niu Z, Hardison M, Person R, Bekheirnia MR, Leduc MS, Kirby A, Pham P, Scull J, Wang M, Ding Y, Plon SE, Lupski JR, Beaudet AL, Gibbs RA, Eng CM. Clinical whole-exome sequencing for the diagnosis of mendelian disorders. N Engl J Med. 2013 Oct 17;369(16):1502-11. doi: 10.1056/NEJMoa1306555. Epub 2013 Oct 2. PMID 24088041
- [Background] Slavotinek A. Clinical care models in the era of next-generation sequencing. Mol Genet Genomic Med. 2016 May 12;4(3):239-42. doi: 10.1002/mgg3.225. eCollection 2016 May. No abstract available. PMID 27247951
- [Derived] Rego S, Hoban H, Outram S, Zamora AN, Chen F, Sahin-Hodoglugil N, Anguiano B, Norstad M, Yip T, Lianoglou B, Sparks TN, Norton ME, Koenig BA, Slavotinek AM, Ackerman SL. Perspectives and preferences regarding genomic secondary findings in underrepresented prenatal and pediatric populations: A mixed-methods approach. Genet Med. 2022 Jun;24(6):1206-1216. doi: 10.1016/j.gim.2022.02.004. Epub 2022 Apr 8. PMID 35396980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited pediatric patients to this study. We aimed to reach 800 pediatric cases in the beginning of the study, and we completed 529 cases at the end.
Pre-assignment Details: This is an exploratory study to define the diagnostic yield of exome sequencing in this pediatric population. All participants were offered the same test and received the same study procedures. There are no arms in this study.
Period: Overall Study
Arm/Group | Whole Exome Sequencing
Started | 529
Completed | 529
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Whole Exome Sequencing: Following consent and collection of standardized phenotypic data, probands and biological parents will undergo WES with variant analysis conducted utilizing primary gene lists based on referring clinical indication. After results provision and follow up 6 months later, diagnostic yield will be assessed as a measure of clinical utility. Those with a positive result (pathogenic or likely pathogenic variant) divided by the total number of cases sequenced will give the diagnostic yield. The assessment will be per pediatric case (proband), meaning, genomic data from biological parents and occasionally from siblings will be used to support the diagnosis for the proband.
  Whole Exome Sequencing: Whole Exome Sequencing is a form of Next Generation Sequencing allowing investigators to assess the coding regions of many thousands of genes to find variants implicated in disease.
Arm/Group | Whole Exome Sequencing
Number analyzed (Participants) | 529
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 525
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 5.0 [0 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239
  Male | 290
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian, Native American, Alaska Native | 5
  Asian | 45
  Black/African American | 19
  Native Hawaiian, Pacific Islander | 5
  White/European American | 99
  Middle Eastern/North African | 22
  Hispanic/Latino(a) | 226
  More than one | 40
  Unknown/none of these fully describe me | 68
Region of Enrollment [Number; unit: participants]
  United States | 529

OUTCOME MEASURES:

1. Primary Outcome: Number of Pediatric Patients With a Positive Exome Sequencing Result
Description: Number of pediatric patients with a diagnostic result among all patients where exome was performed.
  A positive exome sequencing result means the identification of a pathogenic or likely pathogenic gene variant to explain the child's condition.
  The definition of pediatric was expanded to include participants over the age of 18 if they were being followed by UCSF pediatrics department if they were patients at the pediatrics department before they were 18 years old.
Time Frame: At the completion of data collection (follow-up visit at 6-12 months after return of results)
Population: 529 Probands total were enrolled in the study, 525 pediatric participants, and 4 were over the age of 18.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Exome Sequencing
Number analyzed (Participants) | 529
Participants | 142

ADVERSE EVENTS:
Time Frame: Each patient was followed for 6-9 months
Arm/Group | Whole Exome Sequencing
All-Cause Mortality (participants affected / at risk) | 0/529
Serious Adverse Events (participants affected / at risk) | 0/529
Other Adverse Events (participants affected / at risk) | 0/529

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03525431/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03525431/SAP_001.pdf
  • Informed Consent Form (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03525431/ICF_002.pdf